CLINICAL TRIAL: NCT06512051
Title: A Phase IB /II, Multicenter, Open-Label Study of Safety, Tolerability and Efficacy of SHR-A2102 for Injection With Adebrelimab With or Without Other Antitumor Therapy in Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: A Trial of SHR-A2102 With Adebrelimab With or Without Other Antitumor Therapy in Advanced or Metastatic Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A2102-205
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Advanced or Metastatic Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Injections; Cisplatin; Carboplatin; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): SHR-A2102+Adebrelimab+Cisplatin/Carboplatin
  Interventions: Drug: SHR-A2102 for Injection; Drug: Adebrelimab Injection; Drug: Cisplatin injection; Drug: Carboplatin injection
- Treatment group B (Experimental): SHR-A2102+Adebrelimab+Bevacizumab
  Interventions: Drug: SHR-A2102 for Injection; Drug: Adebrelimab Injection; Drug: Bevacizumab Injection

INTERVENTIONS:
Drug: SHR-A2102 for Injection — Drug: SHR-A2102 for injection.
Drug: Adebrelimab Injection — Adebrelimab injection.
Drug: Cisplatin injection — Cisplatin injection.
  Arms: Treatment group A
Drug: Carboplatin injection — Carboplatin injection.
  Arms: Treatment group A
Drug: Bevacizumab Injection — Bevacizumab injection.
  Arms: Treatment group B

SUMMARY:
The study is being conducted to evaluate the safety, tolerability and efficacy of SHR-A2102 with Adebrelimab with or without other Antitumor Therapy in Advanced or Metastatic Non-small cell lung Cancer.

To explore the reasonable dosage of SHR-A2102 for Advanced or Metastatic Non-small cell lung Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to give informed consent, have signed informed and able to comply with the treatment plan to visit the tests and other procedural requirements.
2. The age of signing the informed consent is 18 -70 years, regardless of gender.
3. Provide archived or fresh tumor tissue for vendor test.
4. At least one measurable lesion according to RECIST v1.1 criteria.
5. Patients with locally advanced or metastatic non-small cell lung cancer who have been confirmed by histological or cytological examination to be inoperable and unable to undergo radical radiotherapy or chemotherapy.
6. The ECOG score is 0 or 1.
7. Expected survival ≥12 weeks.
8. Good level of organ function.
9. Male subjects whose partners are women of childbearing age and female subjects who are fertile are required to use highly effective contraceptive methods.

Exclusion Criteria:

1. Active or symptomatic brain metastases.
2. With the exception of patients diagnosed with any other malignancy, except those who have achieved complete remission at least 5 years prior to screening and have ended adjuvant therapy, can be treated locally and have a clear medical record of cure, such as basal cell or squamous cell carcinoma of the skin, superficial bladder cancer in situ, carcinoma in situ of the cervix, breast ductal carcinoma in situ, and papillary carcinoma of the thyroid.
3. Uncontrollable moderate to large amounts of pleural effusion, peritoneal effusion or pericardial effusion.
4. Patients with uncontrolled tumor-related pain .
5. Have antitumor therapy was received 4 weeks before the start of the study.
6. Perform non-chest radiation therapy with >30 Gy within 28 days before dosing, chest radiation therapy with >30 Gy within 24 weeks before first dosing, and radiation therapy with ≤30 Gy within 14 days before first dosing.
7. Subjects who are participating in another clinical study or whose first dose is less than 4 weeks from the end of the previous clinical study (last dose), or the 5 half-life of the investigational drug, whichever is longer.
8. Surgical procedures requiring tracheal intubation and general anesthesia were performed within 28 days prior to the initial study, diagnostic or superficial surgery was performed within 7 days prior to the initial study, or elective surgery was expected during the trial period.
9. Toxicity and/or complications of previous antitumor therapy did not return to NCI-CTCAE level ≤1 or exclusion criteria
10. Systemic immunosuppressive therapy was administered within 14 days prior to the first study.
11. Subjects with a prior history of interstitial pneumonia/non-infectious pneumonia requiring hormone therapy, and currently known or suspected interstitial pneumonia/non-infectious pneumonia.
12. The presence of any active, known or suspected autoimmune disease.
13. Subjects with severe cardiovascular and cerebrovascular diseases.
14. Subjects who had a severe infection within 28 days prior to the first dose
15. Active hepatitis B or active hepatitis C.
16. Patients with active pulmonary tuberculosis within 1 year prior to enrolment.
17. Clinically significant bleeding symptoms or significant bleeding tendency occurred within 1 month before the first medication
18. History of immune deficiency
19. Live attenuated vaccines were used within 28 days prior to initial study administration or during the expected study treatment；
20. Female subjects who are pregnant or plan to become pregnant during the study period.
21. Uncontrollable mental illness and other conditions known to affect the completion of the study process, such as alcohol, drug or substance abuse, and criminal detention.
22. Per the investigator's judgment, there are any other circumstances that may increase the risk of participating in the study, interfere with the study results, or make participation in the study inappropriate.
23. Having a bleeding tendency, a high risk of bleeding, coagulation dysfunction or thrombosis tendency (for patients using bevacizumab).
24. Poorly controlled hypertension (with regular antihypertensive treatment, systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 100 mmHg), as well as previous occurrence of hypertensive crisis or hypertensive encephalopathy (in patients using bevacizumab).
25. Within 6 months prior to the first administration of the medication, had a major vascular disease (for patients using bevacizumab).
26. If within 7 days prior to the first administration of the drug, the patient had used the full dose of oral or injectable anticoagulant or thrombolytic drugs for therapeutic purposes, prophylactic anticoagulation treatment for the open intravenous infusion system is permitted, and prophylactic use of low-molecular-weight heparin (for patients using bevacizumab) is also allowed.
27. Within 7 days prior to the first administration, the patient has used or needs to use aspirin, dipyridamole, ticlopidine, clopidogrel, cilostazol or other drugs that inhibit platelet function (for patients using bevacizumab).
28. Having severe, non-healed wounds, active ulcers or untreated fractures (for patients using bevacizumab).
29. Within 6 months prior to the first administration of the drug, there had been a history of gastrointestinal perforation. During the screening process, clinical symptoms or signs indicated the presence of intestinal obstruction (for patients using bevacizumab).
30. CT/MRI indicated that the tumor surrounded or invaded major blood vessels (for patients who received bevacizumab treatment).
31. Subjects who have previously received systemic treatment with anti-angiogenic drugs such as VEGF/VEGFR inhibitors, including but not limited to bevacizumab, recombinant human endostatin, anlotinib, etc. (patients who used bevacizumab).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
RP2D | through phase IB completion, an average of 1 years
  RP2D will be determined on the basis of evaluation on safety, PK, efficacy data in Phase IB stages；
Incidence and severity of AE(DLT) | from Day1 to 90 days after last dose
  According to NCI-CTCAE v5.0 evaluation criteria from Day 1 to 90 days after last dose；
ORR | 18 months after the last subject was enrolled in the group
  efficacy was assessed every 6 weeks within 48 weeks and every 9 weeks after 48 weeks s as determined by RECIST1.1

SECONDARY OUTCOMES:
DCR | 18 months after the last subject was enrolled in the group
  Since C1D1 every 6 weeks within 48 weeks and every 9 weeks after 48 weeks, and the proportion of subjects whose best response was PR or CR or SD as determined by RECIST1.1；
DOR | 18 months after the last subject was enrolled in the group
  Since C1D1 every 6 weeks within 48 weeks and every 9 weeks after 48 weeks, and the proportion of subjects whose best response was PR or CR or SD as determined by RECIST1.1；
PFS(Investigator evaluation) | 18 months after the last subject was enrolled in the group
  Since C1D1 every 6 weeks within 48 weeks and every 9 weeks after 48 weeks, and the proportion of subjects whose best response was PR or CR or SD as determined by RECIST1.1；
OS(Investigator evaluation) | 18 months after the last subject was enrolled in the group
  Since C1D1 and death from any cause；

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided